CLINICAL TRIAL: NCT03809169
Title: Rapid On-site Evaluation and Use of a Slim Bronchoscope During Peripheral Endobronchial Ultrasonography for the Investigation of Peripheral Pulmonary Lesion - A Randomized Controlled Factorial Trial
Brief Title: Peripheral EBUS With ROSE vs no ROSE; Slim Bronchoscope Without Guide Sheath vs Standard Bronchoscope With Guide Sheath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: McGill University (Other); Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 88888
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Pulmonary Lesions; Lung Cancer
Keywords: peripheral endobronchial ultrasound; radial endobronchial ultrasound; guide sheath; ultrathin bronchoscope; peripheral pulmonary lesion
MeSH Terms: conditions — Lung Neoplasms | interventions — Rapid On-site Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ROSE with guide sheath (Experimental): Patients will undergo pEBUS with a regular size bronchoscope using the guide sheath technique and presence of ROSE
  Interventions: Procedure: Rapid on-site evaluation (ROSE)
- ROSE without guide sheath (Experimental): Patients will undergo pEBUS with a slim bronchoscope combined with a 1.7mm radial probe but no guide sheath and the presence of ROSE.
  Interventions: Procedure: Rapid on-site evaluation (ROSE); Procedure: Slim bronchoscope without a guide sheath
- Guide sheath without ROSE (Experimental): Patients will undergo pEBUS with a regular size bronchoscope using the guide sheath technique but without ROSE.
  Interventions: Procedure: Standard pEBUS with guide sheath
- No guide sheath without ROSE (Experimental): Patients will undergo pEBUS with a slim bronchoscope combined with a 1.7mm radial probe but no the guide sheath an without the presence of ROSE.
  Interventions: Procedure: Slim bronchoscope without a guide sheath

INTERVENTIONS:
Procedure: Rapid on-site evaluation (ROSE) — Pathologist on site for direct evaluation of specimen adequacy
  Arms: ROSE with guide sheath; ROSE without guide sheath
Procedure: Slim bronchoscope without a guide sheath — peripheral endobronchial ultrasound performed with a slim bronchoscope (3.0 mm outer diameter with a 1.7mm channel) combined with a radial ultrasound probe but without the use of a guide sheath.
  Other Names: Ultrathin bronchoscope with pEBUS
  Arms: No guide sheath without ROSE; ROSE without guide sheath
Procedure: Standard pEBUS with guide sheath — Using a flexible bronchoscope with minimal outer diameter of 4.2mm.
  Arms: Guide sheath without ROSE

SUMMARY:
Peripheral pulmonary lesions (PPL) are defined as nodules or masses that are located in the lung periphery; hence cannot be seen via regular bronchoscopy. Due to their location, establishing a pathological diagnosis can be challenging. Investigations of PPL has significantly evolved in the last decade with the development of new technologies such as peripheral endobronchial ultrasound (pEBUS), virtual bronchoscopy and electromagnetic navigational bronchoscopy (ENB). Although these technologies have allowed physicians to safely biopsy previously difficult to access nodules, their sensitivity have been lower than trans-thoracic needle aspiration (TTNA). In fact, the largest registry to date has found a diagnostic yield of pEBUS of 57% compared to 93% for TTNA. However, TTNA caries substantially more procedural risk than pEBUS with a 25% rate of complication vs 2.8% for pEBUS (1, 2). With increased sensitivity, pEBUS could become the procedure of choice for PPL investigation in view of its safety profile. Rapid on-site evaluation of biopsy samples by a cytopathologist (ROSE) allows for direct evaluation of specimen adequacy. By offering real-time feedback to the bronchoscopist about specimen adequacy, the adding of ROSE to pEBUS could lead to an increase in diagnostic yield, allowing for a faster diagnosis of lung cancer and avoiding the need for further diagnostic procedures. Minitiazuration of broncoscopes can also allow navigation to more distal areas of the lung closer to the PPL. While this may also improve diagnostic yield, other technical modification such as the need for smaller sampling instruments and inability to use a guide sheath may have drawbacks.

This study will use a 2 x 2 factorial design to compare diagnostic yield of pEBUS bronchoscopic PPL sampling with vs. without ROSE as well as with a novel "slim" bronchoscope vs. standard bronchoscope. The investigators aim to randomize 208 patients to independently test each hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old
2. Presence of a peripheral pulmonary lesion (PPL) of ≤5cm (mean short-long on axial CT) suspicious for malignancy.
3. The PPL appears radiologically accessible via pEBUS as assessed by an experienced interventional respirologist.
4. Absence of suspicious mediastinal lymphadenopathy on non-invasive staging defined as N1, N2 or N3 nodes ≥1cm on CT or ≥ moderate uptake on PET/CT unless shown to be negative on invasive sampling. Linear EBUS sampling of nodal stations will otherwise be permitted as part of a staging procedure.
5. Clinical decision made by patient and treating physician to proceed to bronchoscopy.

Exclusion Criteria:

1. Other intervention indicated as primary diagnostic procedure (eg: TTNA, surgical lung biopsy, linear EBUS alone, biopsy of extra-thoracic lesion)
2. Location of lesion not amenable to transbronchial needle aspiration sampling as assessed by an experienced interventional respirologist.
3. Contra-indication to pEBUS or bronchoscopy such as: severe pulmonary hypertension (mean pulmonary arterial pressure of ≥25mmHg with evidence of right heart failure), unstable medical condition or uncorrected coagulopathy.
4. Pregnancy
5. Use of electromagnetic or other navigation system (virtual bronchoscopic planning is allowed)
6. Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Peripheral pulmonary lesion diagnostic yield | 1 month

SECONDARY OUTCOMES:
Sensitivity and specificity for malignancy | weeks up to 1 month
Total procedure time | Intraoperative
Sample adequacy for adjunctive testing if lung cancer | 1 month
  Sample adequacy for EGFR mutation analysis, ALK and PDL1 immunohistochemistry.
Extra diagnostic procedure required for final diagnosis. | 6 months up to 1 year
Complications | 48 hours
  Combination of endpoints following chart review, including but not limited to unplanned hospitalization or emergency room visit, hemoptysis, pneumothorax, chest infection, fever or exacerbation of lung disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Tremblay, MDCM, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Health Sciences Centre, Calgary, Alberta
  - Universite Laval, Québec

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data that underlie the results reported in this article (text, tables, figures and appendices) will be shared with researchers who provide a methodologically sound proposal. Other accessible documents will include the study protocol. Beginning 9 months and ending 36 months following article publications, proposals may be submitted to alain.tremblay@ucalgary.ca. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following article publication
Access Criteria: Shared with researchers who will provide a methodologically sound proposal.

REFERENCES:
- [Derived] Vakil E, Fortin M, Gonzalez AV, Samy L, Chee AC, Dumoulin E, Dvorakova M, Hergott CA, Khalil M, Lampron N, MacEachern P, Martel S, Shieh B, Simon M, Soumagne T, Terzic T, Tremblay A. Ultrathin Bronchoscopy With Radial Endobronchial Ultrasound and Rapid On-Site Evaluation for the Diagnosis of Peripheral Pulmonary Lesions: A Multicenter Randomized Controlled Factorial Trial. Chest. 2025 Oct;168(4):1034-1048. doi: 10.1016/j.chest.2025.05.020. Epub 2025 May 24. PMID 40419109